CLINICAL TRIAL: NCT02083874
Title: Cannabidiol (CBD) for the Management of Cannabis Withdrawal: A Phase II Proof of Concept Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Jan Copeland, Professor/Director NCPIC, The University of New South Wales
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCPIC2014001
Record Dates: First submitted 2014-03-06; First posted 2014-03-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Cannabis Use Disorder
Keywords: cannabidiol; CBD; marijuana; withdrawal; treatment
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CBD (Experimental): Open label CBD
  Interventions: Drug: CBD

INTERVENTIONS:
Drug: CBD
  Other Names: No brand names as cannabidiol is not commercially available

SUMMARY:
Single subject repeated measures design of an open label administration of Cannabidiol (CBD) to 5 participants withdrawing from cannabis use in an inpatient setting. 300mg of CBD will be administered once on day 1, twice on days 2-5 and once on day 6. Participants will be discharged on day 7. CBD will be administered orally in capsules.

ELIGIBILITY:
Inclusion Criteria: Participants must be seeking treatment for cannabis use disorder and report having experienced cannabis withdrawal symptoms in past quit attempts (as defined by participants' experiencing 3 or more symptoms after cessation of prolonged cannabis use or continuing use to avoid withdrawal symptoms). They must meet the criteria for a DSMV current cannabis use disorder and test positive to THC on urinary dip stick test on admission. They must be aged 18-65 and speak English.

Exclusion Criteria: The aim is to exclude individuals with concurrent conditions that jeopardise patient safety or confound study data interpretation. These include (a) presence of another substance use disorder, operationalized as (i) more than twice weekly use of an illicit drug in the last 90 days (other than cannabis), (ii) alcohol AUDIT scores of greater than 15, or a current history of alcohol dependence, (iii) substance use treatment in the last 30 days, or (iv) current prescription drug abuse or dependence (benzodiazepines, opioids or psychostimulants); (b) evidence of unstable or severe medical conditions or cognitive or psychiatric impairment (including developmental disorder, schizophrenia or other psychotic disorders) that may prevent participation; (f) known or suspected allergy to propylene glycol, corn oil; (h) women of child bearing age not on a reliable contraceptive or men intending to start a family with one month of trial participation; (i) pregnant or lactating women; (j) not available for follow-up; (k) no access to telephone; or (l) unwillingness to provide written confirmation that they have been informed about, and will comply with, exclusion from driving when receiving medication. Only persons meeting all criteria will be assessed by trial medical officers and research staff as appropriate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Severity of cannabis withdrawal | 7 days
  Reduction of number and severity of withdrawal symptoms including insomnia, anxiety, agitation, restlessness, low mood. This will be assessed using the only validated scale: The Cannabis Withdrawal Scale
Safety of CBD for cannabis withdrawal | 7 days
  Unwanted effects of any nature will be monitored using the reporting protocols employed in similar studies and monitored by senior addiction specialists. Any SAEs will be reported to the TGA as required.

SECONDARY OUTCOMES:
Treatment retention | 7 days
  Retention in inpatient treatment will be assessed against previous studies of cannabis treatment retention and TAU participants in the unit

CONTACTS AND LOCATIONS:
Overall Officials: Martin Weltman, PhD MD, Principal Investigator — Nepean Blue Mountains Local Health District